CLINICAL TRIAL: NCT03278288
Title: Gamified WellWe-intervention to Promote the Health and Wellbeing of Families With Small Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Turku (Other)
Responsible Party: Principal Investigator, Anni Pakarinen, Doctoral candidate, University of Turku
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: WellWeF2017
Record Dates: First submitted 2017-09-05; First posted 2017-09-11 (Actual); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Health Behavior; Healthy
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Intervention Model Description: Two-arm cluster randomized controlled trial and conducted in four municipalities located in the Southwest Finland. The unit of randomization is one cluster, with one municipality with its Child health clinics representing one cluster. Two municipalities with all together eight Child health clinics are randomly allocated into the intervention arm and two municipalities with all together seven Child health clinics are randomly allocated into the control arm.
Who Masked: Participant
Masking Description: Family participants are masked and control group is not aware of the intervention condition. PHN participants are not masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WellWe-Intervention group (Experimental): WellWe-intervention includes the use of WellWe-app to assess the current situation of the wellbeing of the family at home and utilizing these results using WellWe-app during the health visit in Child health clinic.
  Interventions: Device: WellWe-Intervention group
- Usual care group (No Intervention): Usual care includes the filling of normal paper-based questionnaires to assess the current situation of the wellbeing of the family at home and utilizing these results during the normal health visit in Child health clinic.

INTERVENTIONS:
Device: WellWe-Intervention group — Participants (families) allocated to the intervention group get to use WellWe-app before entering to health visit to assess the current situation of their wellbeing and utilizing these results during the health visit. The access to WellWe-app is permitted throughout the data collection period. Participants (PHNs) randomized to the intervention group get standardized two hour WellWe-training, WellWe-handbook and full access to the WellWe-app during the data collection period.
  Arms: WellWe-Intervention group

SUMMARY:
The study evaluates the effectiveness of the WellWe-intervention in promotion of parental self-efficacy for healthy behaviors and mindfulness in parenting from the perspective of families. Aim is also to evaluate the effectiveness of the WellWe-intervention in facilitation of family-centered approach of the health visit in Child health clinic perceived by the families and Public health nurses (PHN). Half of the participants will receive WellWe-intervention and half of the participants will receive usual care.

DETAILED DESCRIPTION:
Families with pre-school aged children attend to regular health visits in Child health clinics on a yearly basis. During the health visits PHNs assess and promote the health and wellbeing of the whole family through health discussions.

In this study we aim to evaluate whether the addition of gamified method into the health discussion promotes healthy behaviors and mindfulness of the families and increases the family-centered approach of health visit compared to the traditional method.

WellWe-intervention includes the use of gamified WellWe app at home and during the health discussion in the Child health clinic. Usual care includes paper-based questionnaires filled by the parents and health discussion using these questionnaires in the Child health clinic.

ELIGIBILITY:
Inclusion Criteria:

* families: Finnish speaking families with 4-year old child and attend into health visit in Child health clinic during data collection period.
* PHNs: a permanent employee in Child health clinic or deputy employee working in Child health clinic during the data collection period.

Exclusion Criteria:

* families: Child is developmentally disabled to participate to the use of WellWe-app with parents.
* PHNs: Deputy employees working in Child health clinic only a short period of time or temporarily.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-05-15 (Actual); Primary Completion 2018-05 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Change in Parental Self-Efficacy for Healthy Dietary and Physical Activity Behaviors in Preschoolers Scale (PDAP) | at baseline, an average of 2 weeks and an average of 4 months
  In this study we use version of the PDAP consisting of 21 items covering contextual circumstances that may either facilitate or impede parental self-efficacy (PSE) for promoting healthy dietary and physical activity behaviors in preschool children. Responses are made on an 11-point Likert scale, with anchors at 0 (not at all confident), 5 (moderately confident), and 10 (completely confident).

SECONDARY OUTCOMES:
Change in Mindfulness In Parenting Questionnaire (MIPQ) | at baseline and an average of 4 months
  In this study we use the version of the MIPQ including 28 items. For each item, parents respond using a four-point Likert-type rating scale: infrequently (1), sometimes (2), often (3), or almost always (4).
Questionnaire on the family-centered approach of the health visit | an average of 2 weeks
  Questionnaire developed for the purpose of the study for families consists of 6 dichotomous questions (yes/no) and one open-ended question. Questionnaire for the PHNs consists of 3 dichotomous questions (yes/no) and 3 items with four-point Likert-type rating scale and one open-ended question.

OTHER OUTCOMES:
Questionnaire on the background information on the family | at baseline
  Questionnaire developed for the study purposes includes questions of the respondent's gender, age, education, occupation, family circumstances.

CONTACTS AND LOCATIONS:
Overall Officials: Anni Pakarinen, MHSc, Principal Investigator — University of Turku, Finland
Locations (1):
- Child health clinics, Four Municipalities, Southwest Finland, Finland